CLINICAL TRIAL: NCT05358886
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study of BPN14770 in Male Adults (Aged 18 to 45) With Fragile X Syndrome
Brief Title: A Study of BPN14770 in Male Adults (Aged 18 to 45) With Fragile X Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPN14770-CNS-301
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Fragile X Syndrome
Keywords: FXS
MeSH Terms: conditions — Fragile X Syndrome | interventions — BPN14770

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug (Active Comparator): 25mg BID BPN14770
  Interventions: Drug: BPN14770/ zatolmilast
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BPN14770/ zatolmilast — 25mg BID BPN14770
  Arms: Study Drug
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Parallel Group Study of BPN14770 in Male Adults (Aged 18 to 45) with Fragile X Syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Male subject aged 18 to 45 years at screening visit.
2. Subject has FXS with a molecular genetic confirmation of the full fragile X mental retardation-1 (FMR1)mutation (≥200 CGG repetitions).
3. Subject is able to swallow capsules.
4. Current treatment with ≤3 prescribed psychotropic medications. Anti-epileptic medications are permitted and are not counted as psychotropic medications if they are used for the treatment of seizures. Anti-epileptics for other indications, such as the treatment of mood disorders, count towards the limit of permitted medications.
5. Permitted concomitant psychotropic medications must be at a stable dose and dosing regimen for at least 4 weeks prior to screening and must remain stable during the period between screening and the commencement of the study treatment.
6. Anti-epileptic medications must be at a stable dose and dosing regimen for 12 weeks prior to screening and must remain stable during the period between screening and commencement of the study treatment.
7. Subjects with a history of seizure disorder who are currently receiving treatment with anti-epileptics must have been seizure free for 3 months preceding screening or must be seizure free for 2 years if not currently receiving anti-epileptics.
8. Behavioral and other non-pharmacological treatments/interventions must be stable for 4 weeks prior to screening and must remain stable during the period between screening and first dose of study treatment and throughout the study. Minor changes in hours or times of therapy that are not considered clinically significant will not be exclusionary. Changes in therapies provided through a program (eg, due to a vacation) are allowed.
9. Subject must be willing to practice barrier methods of contraception while on the study if sexually active. Abstinence is also considered a reasonable form of birth control in this study population.
10. Subject has a parent, legal authorized guardian, or consistent caregiver.
11. Subject and caregiver are able to attend the clinic regularly and reliably.
12. If subject is his own legal guardian, he is able to understand and sign informed consent to participate in the study.
13. For subjects who are not their own legal guardian, subject's parent/legally authorized guardian is able to understand and sign an informed consent form for their child to participate in the study.
14. If subject is not his own legal guardian, subject must provide assent for participation in the study if he has the cognitive ability to do so.

Exclusion Criteria:

1. Inability to successfully complete the NIH-TCB picture vocabulary and oral reading assessments at screening and baseline. The ability to complete the NIH-TBC oral reading and picture vocabulary subtest at baseline is defined as the ability to complete both subtests, with (1) confirmation from the clinician administering that the test administrations are valid (noted on the administration form) and (2) generation of valid test scores for each test.
2. History of or current cardiovascular, renal, hepatic, respiratory, gastrointestinal, psychiatric, neurologic, cerebrovascular, or other systemic disease that would place the subject at risk or potentially interfere with the interpretation of the safety, tolerability, or efficacy of the study treatment.

   a. Common conditions such as mild hypertension, etc. are allowed per the principal investigator's judgement as long as they are stable and controlled by medical therapy that is constant for at least 4 weeks before randomization.
3. Renal impairment, defined as serum creatinine > 1.25 × ULN at screening
4. Hepatic impairment, defined as ALT or AST elevation > 2 × ULN at screening. Note: LFTs may be repeated after 1 week to evaluate return to acceptable limits; if LFTs remain elevated, the subject is ineligible to participate.
5. Clinically significant abnormalities, in the investigator's judgement, in safety laboratory tests, vital signs, or ECG, as measured during screening.
6. History of substance abuse within the past year, according to investigator assessment.
7. Positive COVID-19 test during screening.
8. Significant hearing or visual impairment that may affect the subject's ability to complete the test procedures.
9. Concurrent major psychiatric condition (eg, major depressive disorder, schizophrenia, or bipolar disorder) as diagnosed by the investigator. Subjects with the additional diagnosis of autism spectrum disorder or anxiety disorder will be allowed.
10. Subject has active diseases that would interfere with participation, such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.
11. Subject is planning to commence psychotherapy or cognitive behavior therapy during the period of the study or had begun psychotherapy or cognitive behavior therapy within 4 weeks prior to screening.
12. Subject is an immediate family member of anyone employed by the sponsor, investigator, or study staff.
13. Subject has a body mass index of less than 18 kg/m2 or greater than 36 kg/m2.
14. Subject has participated in another clinical trial within the 30 days preceding Screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 171 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Toolbox Cognitive Battery cognition crystallized composite score (NIH-TCB CCC) | 13 Weeks
  National Institutes of Health Toolbox Cognitive Battery cognition crystallized composite score (NIH-TCB CCC), which is calculated from the Picture Vocabulary and Oral Reading domains.

SECONDARY OUTCOMES:
Numerical rating scale (NRS) scores based on subject-specific behaviors vs baseline | 13 Weeks
  Numerical rating scale (NRS) scores based on subject-specific behaviors within the domains of Daily Function and Language
Caregiver Global Impression of Improvement (CaGI-I) | 13 Weeks
  Caregiver Global Impression of Improvement (CaGI-I) for the general domains of Daily Function and Language
Clinical Global Impression Improvement (CGI-I) for - Investigator | 13 Weeks
  Clinical Global Impression Improvement (CGI-I) for - Investigator rated the general domains of Daily Function and Language
Vineland-3 Adaptive Behavior Scale (Vineland-3) | 13 Weeks
  Vineland-3 Adaptive Behavior Scale (Vineland-3), using the composite score and domain scores from communication, daily living skills, and socialization
Verbal Knowledge test from the Stanford-Binet (ed 5) (SB-5)IQ | 13 Weeks
  Verbal Knowledge test from the Stanford-Binet (ed 5) (SB-5) IQ assessment
NIH-TCB domains of Picture Sequence Memory, Flanker Inhibitory Control and Attention, List Sorting Working Memory, Dimensional Change Card Sort, and Speeded Matching | 13 Weeks
  NIH-TCB domains of Picture Sequence Memory, Flanker Inhibitory Control and Attention, List Sorting Working Memory, Dimensional Change Card Sort, and Speeded Matching
Aberrant Behavior Checklist (ABC) scores | 13 Weeks
  Aberrant Behavior Checklist (ABC) scores
Anxiety, Depression, and Mood Scale (ADAMS) scores | 13 Weeks
  Anxiety, Depression, and Mood Scale (ADAMS) scores

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, MD, Principal Investigator — Rush Medical Center
Locations (17):
- United States (17):
  - Amnova Clinical Research, Irvine, California
  - Thompson Autism & Neurodevelopment Center - CHOC, Orange, California
  - UC Davis Health System, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Icahn School of Medicine at Mount Sinai Hospital, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Clinic for Special Children, Strasburg, Pennsylvania
  - Greenwood Genetic Center, Greenville, South Carolina
  - University of Utah and Primary Childrens Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No